CLINICAL TRIAL: NCT07206290
Title: Albuminuria Reduction Trial and Investigation With Survodutide Treatment in CKD
Brief Title: Albuminuria Reduction Study With Survodutide Treatment in Kidney Disease
Acronym: ARTIST-CKD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22774; 2025-523184-37-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-08

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — BI 456906

STUDY DESIGN:
Intervention Model Description: This is a parallel, randomized, double-blind, placebo-controlled clinical trial conducted in 4 countries (Netherlands, Germany, Spain and Australia)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Survodutide (Experimental): 2:1 fashion to a 16 weeks up-titration phase of survodutide (0.3 mg, 0.6 mg, 1.2 mg, 2.4 mg and 3.6 mg subcutaneous injection weekly) followed by a 20 weeks maintenance phase of survodutide s.c. 3.6 mg once weekly
  Interventions: Drug: Survodutide (BI 456906)
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Survodutide (BI 456906) — 0.3 mg, 0.6 mg, 1.2 mg, 2.4 mg, 3.6 mg s.c. weekly
  Arms: Survodutide
Drug: Placebo — Placebo matching survodutide
  Arms: Placebo

SUMMARY:
The ARTIST-CKD trial is a clinical study evaluating the effect of weekly subcutaneous administration of survodutide (3.6 mg) on kidney function in patients with chronic kidney disease (CKD) and elevated albuminuria. The primary objective is to determine whether survodutide leads to early, sustained, and clinically meaningful reductions in albuminuria, regardless of diabetes status.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* eGFR ≥20 and <90 mL/min/1.73m2
* Urinary albumin to creatinine ratio >30 mg/g and <3500 mg/g
* BMI >21 kg/m2
* Stable kidney function (no more than 30% change in eGFR in the 3 months prior to enrolment)
* On a stable maximum tolerated dose of an ACEi/ARB for at least 4 weeks prior to enrolment
* If using an SGLT2 inhibitor, receiving a stable dose for at least 8 weeks prior to enrolment
* Willing to sign an informed consent

Exclusion Criteria:

* Diagnosis of type 1 diabetes
* Cardiovascular event within 3 months prior to enrolment
* Treatment with GLP-1RA for <12 weeks prior to screening
* Evidence of severe hepatic impairment determined by any one of: ALT or AST values exceeding 3x ULN, a history of hepatic encephalopathy, a history of oesophageal varices, or a history of portocaval shunt;
* Active pregnancy or breastfeeding
* History of kidney or liver transplant
* Active malignancy
* Suggestive evidence of adrenal insufficiency
* Acute pancreatitis <180 days prior to screening
* History of chronic pancreatitis or idiopathic acute pancreatitisPersonal or family history of multiple endocrine neoplasia type 2 (MEN2) or familial medullary thyroid carcinoma
* Calcitonin levels ≥100 pg/mL or 29.26 pmol/L
* Personal history of non-familial medullary thyroid carcinoma
* History of severe hypersensitivity or contraindications to any glucagon RA or GLP-1 RA
* Uncontrolled arterial hypertension (mean semi supine systolic blood pressure (SBP) ≥180 mmHg or diastolic blood pressure (DBP) ≥110 mmHg)
* Any medication, surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of medications including, but not limited to any of the following:

  * History of active inflammatory bowel disease within the 6 months;
  * Major gastrointestinal tract surgery as determined by the physician;
  * Pancreatitis within 6 months.
  * GI ulcers and/or bleeding within 6 months;
  * Evidence of urinary obstruction or difficulty in voiding at screening.
* Participation in any clinical trial within 3 months prior to initial dosing.
* Donation or loss of ≧400 ml blood within 8 weeks prior to initial dosing.
* History of drug or alcohol abuse within the 12 months prior to dosing, or evidence of such abuse as indicated by the laboratory assays conducted during the screening or according to investigator's assessment.
* History of noncompliance to medical regimens or unwillingness to comply with the study protocol.
* Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study.
* Women of childbearing potential (WOCBP):

  * WOCBP who are unwilling or unable to use an acceptable method of contraception to avoid pregnancy throughout the study and for up to 8 weeks after the last dose of study drug in such a manner the risk of pregnancy is minimized.
  * WOCBP must have a negative serum or urine pregnancy test result (minimum sensitivity 25 IU/L or equivalent of HCG) at screening.
* Vulnerable (i.e. under guardianship) or mentally incapacitated subjects (i.e. not able to understand and sign the informed consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in first morning void UACR | From baseline to week 32/36
  Average of first morning void urine samples collected at week 32 and 36 will be used to decrease random day-to-day variability and increase precision (and statistical power).

SECONDARY OUTCOMES:
eGFR (creatinine, cystatin C, and creatinine-cystatin C) | From baseline to week 36
Iohexol measured GFR | From baseline to week 36
  Subset of 60 participants
UACR and eGFR during 4-week wash-out | From week 36 to 40
Perirenal and renal sinus fat measured by MRI | From baseline to week 36
  Same subset of 60 participants with Iohexol GFR
Subcutaneous and visceral fat assessed by MRI | From baseline to week 36
  Same subset of 60 participants with Iohexol GFR
Body weight | From baseline to week 36
Waist circumference | From baseline to week 36
Systolic and diastolic blood pressure | From baseline to week 36

OTHER OUTCOMES:
HbA1c | From baseline to week 36
High-sensitivity C-reactive protein | From baseline to week 36
NT-proBNP | From baseline to week 36
Renal blood flow measured by MRI | From baseline to week 36
  Same subset of 60 participants with Iohexol GFR

IPD SHARING:
Plan to Share IPD: No